CLINICAL TRIAL: NCT07385846
Title: Pilot Study for the Use of Navigated Focused Ultrasound and Pembrolizumab in the Treatment of Recurrent WHO Grade 4 IDH-Wildtype Glioblastoma With Mismatch Repair Deficiency: A Phase I Clinical Trial
Brief Title: Pilot Study of Navigated Focused Ultrasound and Pembrolizumab in the Treatment of Recurrent WHO Grade 4 IDH-Wildtype Glioblastoma With Mismatch Repair Deficiency
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jennifer Leddon (Other)
Collaborators: NaviFUS Corporation (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Leddon, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCC-BN-25-02
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma; Mismatch Repair Deficiency
MeSH Terms: conditions — Glioblastoma; Turcot syndrome | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: In this phase I clinical trial, 6-8 patients with recurrent glioblastoma and identified mismatch repair (MMR) deficiency will be administered pembrolizumab along with focused ultrasound sonication following surgery for recurrent glioblastoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Pembrolizumab + focused ultrasound sonication (Experimental): Pembrolizumab along with focused ultrasound sonication following surgery for recurrent glioblastoma. Treatment dosing will be 200mg of pembrolizumab every three weeks for up to six months or until disease progression, whichever occurs first. The primary endpoint will be safety and tolerability, with secondary efficacy endpoints and exploratory biomarker and radiographic analyses.
  Interventions: Drug: Pembrolizumab; Device: Navifus Focused Ultrasound Sonification

INTERVENTIONS:
Drug: Pembrolizumab — Treatment dosing will be 200mg of pembrolizumab every three weeks for up to six months or until disease progression, whichever occurs first.
Device: Navifus Focused Ultrasound Sonification — Focused Ultrasound Sonification- Post Pembro infusion, patients will received NaviFUS sonication to the complete volume of the tumor resection bed (as limited by anatomic constraints relative to the tumor extension) following microbubble (Bracco Imaging, SonoVue® or Lumason®; 0.1 mL/Kg; maximum 4.8 mL) administration on a 2-minute schedule. The NaviFUS procedure will be guided using the compatible navigation system, Medtronic StealthStation®. Microbubble administration and operation of the NaviFUS unit will be completed by qualified delegated study investigators. Treatment sessions will occur every 3 weeks for 6 months or until evidence of disease progression, whichever occurs first. A 6-month treatment duration was determined in order to report a 6-month PFS rate as one of the secondary outcomes for this study population.

SUMMARY:
Navigated Focused Ultrasound and Pembrolizumab in the Treatment of Recurrent WHO Grade 4 IDH-Wildtype Glioblastoma with Mismatch Repair Deficiency.

DETAILED DESCRIPTION:
In this phase I clinical trial, 6-8 patients with recurrent glioblastoma and identified mismatch repair (MMR) deficiency will be administered pembrolizumab along with focused ultrasound sonication following surgery for recurrent glioblastoma. Treatment dosing will be 200mg of pembrolizumab every three weeks for up to six months or until disease progression, whichever occurs first. The primary endpoint will be safety and tolerability, with secondary efficacy endpoints and exploratory biomarker and radiographic analyses

ELIGIBILITY:
Inclusion Criteria:

1. Patient previously diagnosed with WHO grade 4 IDH-wildtype GBM, determined through genomic and/or histopathological analysis.
2. Prior treatment for GBM with surgical resection and standard of care TMZ and radiation therapy.
3. Patient who has undergone repeat surgery (including biopsy or resection) for rGBM.
4. MMR deficiencies confirmed per standard of care immunohistochemical analysis or Next Generation Sequencing (NGS) of the patient's surgical sample from the time of initial GBM diagnosis or recurrence.
5. Area of sonication using the NaviFUS platform is >30 mm from the skull surface, assessed on the Investigator's review of the screening MRI.
6. Age ≥18 years.
7. Karnofsky Performance Scale (KPS) >70.
8. Adequate organ and marrow function:

   Leukocytes ≥2,500/mm3 Absolute Neutrophil Count ≥1,500/mm3 Absolute Lymphocyte Count ≥800/mm3 Platelets ≥100,000/mm3 Hemoglobin ≥8 g/dL
9. Negative serum or urine pregnancy test in a female patient of childbearing potential.
10. Patient or a legally-authorized representative must provide study-specific informed consent.

Exclusion Criteria:

1. Multifocal or leptomeningeal disease observed at the time of GBM recurrence.
2. Patient for whom the repeat surgical cavity is ≤30 mm from the skull surface or otherwise not reasonably accessible for sonification using the NaviFUS platform, assessed on screening MRI.
3. Patient with a prior or concurrent malignancy that is deemed to be clinically significant in the context of rGBM.
4. Patient receiving concurrent treatment with an immune checkpoint inhibitor, other investigational agent, or live vaccine administered within 14 days prior to the first dose of trial treatment.
5. Prior treatment with an immune checkpoint inhibitor agent.
6. Period of less than 28 days from the time of the patient's receipt of other systemic anti-cancer therapies to the proposed date of first trial treatment.
7. Treatment with systemic corticosteroids at an increased dose or dose of ≥10 mg of prednisone (or equivalent) daily within the 5 days prior to starting trial treatment, or treatment with systemic corticosteroids for other indications.
8. Patient with a history of organ transplant or autoimmune disorder requiring active immunosuppression.
9. Patient with current recreational drug use or a history of substance use disorder.
10. Patient with an active concurrent comorbidity that, in the opinion of the Investigator, would pose a safety concern for the patient's participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety of using navigated focused ultrasound (NaviFUS) CTCAE v6.0 | Assessed at each study visit from baseline through 2 years.
  To evaluate the safety of using navigated focused ultrasound (NaviFUS) combined with pembrolizumab (PEM) after repeat surgery for patients with recurrent glioblastoma (rGBM) and mismatch repair (MMR) deficiency. Given that NaviFUS and PEM have defined intracranial dosing, no dose-escalation scheme will be employed. A CTCAE v6.0 grade 4 or higher toxicity probably or definitely attributable (see Section 13.2.3) to the administration of NaviFUS or PEM will be used as the definition for unacceptable toxicity
Feasibility of using navigated focused ultrasound (NaviFUS) -CTCAE v6.0 criteria | Assessed at each study visit from baseline through 2 years.
  To evaluate feasibility of using navigated focused ultrasound (NaviFUS) combined with pembrolizumab (PEM) after repeat surgery for patients with recurrent glioblastoma (rGBM) and mismatch repair (MMR) deficiency. Given that NaviFUS and PEM have defined intracranial dosing, no dose-escalation scheme will be employed. A CTCAE v6.0 grade 4 or higher toxicity probably or definitely attributable (see Section 13.2.3) to the administration of NaviFUS or PEM will be used as the definition for unacceptable toxicity

SECONDARY OUTCOMES:
Overall survival- standard Kaplan-Meier method and calculated from the date of GBM diagnosis | Baseline through 2 years
  To evaluate overall survival (OS) in patients treated with NaviFUS combined with PEM after repeat surgery for patients with rGBM and MMR deficiency.
Progression free survival - standard Kaplan-Meier method and calculated from the date of GBM diagnosis | Baseline through 2 years
  To evaluate progression free survival (PFS) in patients treated with NaviFUS combined with PEM after repeat surgery for patients with rGBM and MMR deficiency.

OTHER OUTCOMES:
Baseline levels of markers of immune function and genetic repair | Baseline
  To evaluate levels of baseline tumor markers related to immune and genetic repair function, including PD-L1, microsatellite instability (MSI), and tumor mutational burden (TMB).
radiographic response to treatment in patients with postsurgical residual disease as determined via mRANO criteria | Baseline
  To evaluate radiographic treatment response according to Modified Response Assessment in Neuro-Oncology (mRANO) criteria prior to treatment with NaviFUS combined with PEM in patients with postsurgical residual tumor.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided